CLINICAL TRIAL: NCT00977275
Title: The Treatment of T1N0 Invasive Breast Carcinoma by Local Excision and Interstitial Implant
Brief Title: Treatment of T1N0 Invasive Breast Carcinoma by Local Excision Implant
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Alphonse Taghian, MD, PhD, Chief Breast Radiation Oncology, MGH, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 97-585
Record Dates: First submitted 2009-09-11; First posted 2009-09-15 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Breast Cancer
Keywords: early stage invasive breast cancer; Partial breast irradiation; interstitial implant
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Radiation: Interstitial Implant Brachytherapy — Via tubes placed at the time of wide local excision delivered over 5 days

SUMMARY:
The purpose of this study is to evaluate radiation therapy directed to a small region of the breast in women who were recently diagnosed with early stage invasive breast cancer.

DETAILED DESCRIPTION:
* When participants undergo surgery to remove the tumor (lumpectomy), it will be followed by the placement of small flexible tubes throughout the region surrounding the site of operation. These tubes will remain in place for 7-9 days following the surgery.
* The first 2-3 days, the tubes will not contain radioactivity. This time is used to do all the calculations necessary for treatment and to check the findings in the breast tissue that was removed. After 2-3 days, the tubes will be filled with a radioactive wire which will remain in place for the next 5 days. During this period of time, participants will be required to remain within the hospital. At the end of these 5 days, the radioactive wires and tubes will be removed.

ELIGIBILITY:
Inclusion Criteria:

* Low risk of multifocal disease within the breast whose tumor location is favorable for brachytherapy catheter placement
* Diagnosis of invasive breast carcinoma (biopsy or fine needle aspiration cytology) and be clinical stage T1N0 (primary tumor < 2cm, clinically negative nodes)
* Location of primary tumor is not immediately adjacent to the nipple of chest wall
* No evidence of two or more separate tumors within the breast
* All histologic types and pathologic grades of primary tumor
* No extensive intraductal component (substantial intraductal carcinoma away from the primary tumor location)
* No lymphatic or vascular invasion
* Lymph node staging by sentinel node excision or axillary dissection confirms node negative status (If node positive, implant is used to deliver boost to tumor bed)
* Assessment of final surgical margins should be predominantly negative, but a single small region of focal positivity is allowable as it is for whole breast radiation
* 18 years of age or older

Exclusion Criteria:

* Tumor is too close to the chest wall to allow placement of catheters
* Contraindications to radiation therapy are present, including a history of scleroderma, systemic lupus or other active connective tissue disease, pregnancy, or prior chest wall radiation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 1997-06; Primary Completion 2006-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
To determine if interstitial implant brachytherapy to radical radiation doses is feasible following wide local excision of T1N0 breast carcinoma | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Alphonse Taghian, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Result] Hattangadi JA, Powell SN, MacDonald SM, Mauceri T, Ancukiewicz M, Freer P, Lawenda B, Alm El-Din MA, Gadd MA, Smith BL, Taghian AG. Accelerated partial breast irradiation with low-dose-rate interstitial implant brachytherapy after wide local excision: 12-year outcomes from a prospective trial. Int J Radiat Oncol Biol Phys. 2012 Jul 1;83(3):791-800. doi: 10.1016/j.ijrobp.2011.09.003. Epub 2011 Nov 16. PMID 22099046
- [Result] Lawenda BD, Taghian AG, Kachnic LA, Hamdi H, Smith BL, Gadd MA, Mauceri T, Powell SN. Dose-volume analysis of radiotherapy for T1N0 invasive breast cancer treated by local excision and partial breast irradiation by low-dose-rate interstitial implant. Int J Radiat Oncol Biol Phys. 2003 Jul 1;56(3):671-80. doi: 10.1016/s0360-3016(03)00071-3. PMID 12788172